CLINICAL TRIAL: NCT03977896
Title: Pilot Study to Evaluate the Feasibility of Hybrid Brain Imaging 11C-MET PET/MRI of Posterior Brain Fossa Tumors in Children
Brief Title: Feasibility of 11C-MET PET/MRI Imaging in Pediatric Brain Fossa Tumors
Acronym: TI-TFCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0867
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Posterior Brain Fossa Tumors in Children
Keywords: PET/MRI; 11C-MET; posterior brain fossa tumors; children; surgery; feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 11C-MET PET/MRI (Experimental)
  Interventions: Procedure: 11C-MET PET/MRI

INTERVENTIONS:
Procedure: 11C-MET PET/MRI — Except PET/MRI imaging, all the examinations will be done according to the patient's usual care.
  PET/MRI imaging will be realized within max 7 days after children enrollment, and the surgery (usual care) will be performed within max 4 days after PET/MRI imaging.
  PET/MRI imaging will include the following sequences: T1axial, Diffusion, Magnetic susceptibility post-Gadolinium injection, 3DT1 pre and post-Gadolinium injection, and Arterial Spin Labelling Imaging (ASL).

SUMMARY:
Brain tumors are the most common solid tumors in children and are the second most common cause of cancer-related death among this population. Posterior brain fossa tumors represent about 50% of children brain tumors.

Recently, knowledge in molecular biology has permitted to identify different tumors subgroups of very different prognosis. Today, surgery removal of the tumor is the mandatory. Neuro-oncological treatment differs depending on the histological and molecular subgroup. With classical Magnetic Resonance Imaging (cMRI), distinction between different types of posterior fossa tumors remains difficult.

Positron Emission Tomography combined with MRI (PET/MRI) has proven its benefits for the management of brain tumors. The direct spatiotemporal correlation makes possible the assessment of metabolic, anatomical and functional information. PET/MRI would provide precisions on the pre-therapeutic characterization of tumors, which could permit to modify the patients' care.

L- [methyl-11C] methionine (11C-MET) is currently the gold-standard tracer used in neuro-oncology, but few data exists in children. 11C-MET PET/MRI assessment seems promising, but has not been studied enough. To the best of our knowledge, there is no specific study on primary brain tumors of the posterior fossa in children using 11C-MET PET/MRI.

The primary objectives of this first pilot study is to evaluate the practical feasibility of 11C-MET PET/MRI imaging (machine accessibility and imaging interpretability) before surgery in a population of children older than 5 years old with posterior fossa tumors.

The secondary objectives aim to describe :

* the PET/MRI parameters of the different tumors studied,
* and the patient's participation acceptation.

This feasibility study will allow us to standardize the PET/MRI measurements; this could allow us to discriminate, in a larger study, the different tumor subgroups before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 5 years old and < 18 years old at enrollment,
* with primary posterior brain fossa tumor, metastatic or not,
* hospitalized in the Department of Pediatric Neurosurgery of Femme-Mère-Enfant Hospital, and for whom a surgery is scheduled,
* covered by national health insurance,
* patient's parents or legal guardians who have provided written informed consent prior to participation in the study.

Exclusion Criteria:

* Patients with contraindication for MRI (claustrophobia, carrying metallic object)
* Patients with contraindication for Gadolinium injection (including pregnancy and breastfeeding)
* patient with recurring posterior brain fossa tumor
* patient with brain stem infiltrative tumor

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
number of patients who performed the PET/MRI | 7 days
number of patients called in for PET/MRI who have not realized the PET/MRI | 7 days
number of patients with good quality of the imaging | 7 days
  The interpretability of the imaging will be evaluated by a Review Committee (two pairs composed each by a radiologist (for MRI imaging) and a nuclear physician (for PET imaging)). The imaging will be classified under good or bad quality

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Aurélien BEURIAT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Groupement Hospitalier Est - Hôpital Femme Mère Enfant - Service de Neurochirurgie Pédiatrique, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beuriat PA, Flaus A, Portefaix A, Szathmari A, Janier M, Hermier M, Lorthois-Ninou S, Scheiber C, Isal S, Costes N, Merida I, Lancelot S, Vasiljevic A, Leblond P, Faure Conter C, Saunier C, Kassai B, Vinchon M, Di Rocco F, Mottolese C. Preoperative 11 C-Methionine PET-MRI in Pediatric Infratentorial Tumors. Clin Nucl Med. 2024 May 1;49(5):381-386. doi: 10.1097/RLU.0000000000005174. Epub 2024 Mar 15. PMID 38498623